CLINICAL TRIAL: NCT06238089
Title: A Novel Way to Understand and Communicate the Burden of Antipsychotic Prescribing for Adults Across Specialist Intellectual Disability Services in England and Wales.
Brief Title: Anti-psychotic Drug Prescribing Patterns Within Specialist Adult ID Services in England and Wales
Acronym: APHID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Professor Rohit Shankar, Professor in Neuropsychiatry, University of Plymouth
Other Study IDs: 4548; TRUST/VC/AC/SG/6328-9580 (Other Grant/Funding Number: The Baily Thomas Charitable Fund); 331470 (Other: IRAS)
Record Dates: First submitted 2024-01-10; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Intellectual Disability
Keywords: Intellectual Disability; Learning Disability; Anti-psychotic treatments; Over-prescribing; Psychotropic
MeSH Terms: conditions — Intellectual Disability; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Eligible patients who have had a psychiatric review by specialist adult ID services in 2017.: Adults with an intellectual disability who are under the care of ID services in receipt of >2 oral and/or long-acting intra-muscular (IM) injectable anti-psychotic treatments (depots), who have had a psychiatric review by specialist adult ID services in 2017.
- Eligible patients who have had a psychiatric review by specialist adult ID services in 2018.: Adults with an intellectual disability who are under the care of ID services in receipt of >2 oral and/or long-acting IM injectable anti-psychotic treatments (depots), who have had a psychiatric review by specialist adult ID services in 2018.
- Eligible patients who have had a psychiatric review by specialist adult ID services in 2019.: Adults with an intellectual disability who are under the care of ID services in receipt of >2 oral and/or long-acting IM injectable anti-psychotic treatments (depots), who have had a psychiatric review by specialist adult ID services in 2019.
- Eligible patients who have had a psychiatric review by specialist adult ID services in 2020.: Adults with an intellectual disability who are under the care of ID services in receipt of >2 oral and/or long-acting IM injectable anti-psychotic treatments (depots), who have had a psychiatric review by specialist adult ID services in 2020.
- Eligible patients who have had a psychiatric review by specialist adult ID services in 2021.: Adults with an intellectual disability who are under the care of ID services in receipt of >2 oral and/or long-acting IM injectable anti-psychotic treatments (depots), who have had a psychiatric review by specialist adult ID services in 2021.
- Eligible patients who have had a psychiatric review by specialist adult ID services in 2022.: Adults with an intellectual disability who are under the care of ID services in receipt of >2 oral and/or long-acting IM injectable anti-psychotic treatments (depots), who have had a psychiatric review by specialist adult ID services in 2022.
- Eligible patients who have had a psychiatric review by specialist adult ID services in 2023.: Adults with an intellectual disability who are under the care of ID services in receipt of >2 oral and/or long-acting IM injectable anti-psychotic treatments (depots), who have had a psychiatric review by specialist adult ID services in 2023.

SUMMARY:
The overall aim of this observational study is to establish the anti-psychotic prescribing patterns across specialist intellectual disability (ID) services in England and Wales by collecting cross-sectional retrospective data at 7 annual time-points (1st July) from 2017 to 2023.

DETAILED DESCRIPTION:
Feasibility protocol objectives:

1. Is it feasible to identify People with Intellectual Disabilities (PwID) who have been prescribed 2 or more anti-psychotic medications over 7 years retrospectively.
2. It is possible to obtain a complete data set for each patient identified and therefore be able to explore the prescribing patterns across the eight sites.
3. Is it feasible to quantify anti-psychotic treatment (APT) prescribing in PwID as chlorpromazine equivalent dose values across different healthcare Trusts in England and Wales.

   Main objectives:
4. To explore yearly and overall prescribing patterns among PwID (with or without mental-health reasons (psychiatric co-morbidities)) in receipt of ≥2 forms of anti-psychotic treatment (multiple) over time?
5. How has multiple anti-psychotic treatment prescribing changed between 2017 and 2023 using chlorpromazine equivalent dose values, in PwID with mental health and no mental health indications?
6. What has been the impact of the COVID-19 pandemic (and corresponding lockdown restrictions in England and Wales) on multiple anti-psychotic treatment prescribing among PwID?
7. Can the NHS England Statistical Process Control tool (SPC) be utilised to track yearly anti-psychotic treatment prescribing among PwID receiving multiple forms of anti-psychotic treatment, and monitor variation between services (sites) and patient groups (e.g. psychiatric co-morbidities; challenging behaviour).

ELIGIBILITY:
Inclusion Criteria:

* Patient had psychiatric review by specialist adult ID services in the last year (e.g. for a patient to be included at 1st June 2017, data to be recorded from the most recent psychiatric review within the period between 1st January 2017 - 31st December 2017).
* Patient has a diagnosis of ID
* Patient under the care of specialist adult ID services
* Patient on >2 anti-psychotic treatments (oral and IM injectable (depots))

Exclusion Criteria:

* Patients treated with Clozapine
* Under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Intellectual Disabilities under the care of ID services in receipt of >2 oral and/or long-acting IM injectable anti-psychotic treatments (depots).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The differences in chlorpromazine equivalent dose values in PwID prescribed multiple anti-psychotic treatment across the 7-annual timepoints and across the 8 sites. | 2017-2023
  Main objective: To explore yearly and overall prescribing patterns among PwID (with or without mental-health reasons (psychiatric co-morbidities)) in receipt of ≥2 forms of anti-psychotic treatment (multiple) over time.
The differences in chlorpromazine equivalent dose values in PwID prescribed multiple anti-psychotic treatment, with mental health indications, compared to those with no mental health indications between 2017 and 2023. | 2017-2023
  Main objective: How has multiple anti-psychotic treatment prescribing changed between 2017 and 2023 using chlorpromazine equivalent dose values, in PwID with mental health and no mental health indications?
The differences in chlorpromazine equivalent dose values in PwID prescribed multiple anti-psychotic treatment before, during and after the COVID-19 pandemic. | 2017-2023
  Main objective: What has been the impact of the COVID-19 pandemic (and corresponding lockdown restrictions in England and Wales) on multiple anti-psychotic treatment prescribing among PwID?
SPC will be used to compare trends in multiple APT prescribing within/across participating healthcare trusts and utilised to track yearly oral/depots anti-psychotic treatment prescribing and monitor variation between services & patient groups. | 2017-2023
  Main objective: Can the SPC be utilised to track yearly anti-psychotic treatment prescribing among PwID receiving multiple forms of anti-psychotic treatment, and monitor variation between services (sites) and patient groups (e.g. psychiatric co-morbidities; challenging behaviour)?

OTHER OUTCOMES:
Number (%) of PwID successfully identified who have been prescribed more than 2 anti-psychotic medications yearly over 7. | Through study completion, an average of 6 months
  Feasibility objective: Is it feasible to identify PwID who have been prescribed 2 or more anti-psychotic medications over 7 years retrospectively?
Number (%) of PwID with a complete data set. | Through study completion, an average of 6 months
  Feasibility objective: Is it possible to obtain a complete data set for each patient identified and therefore be able to explore the prescribing patterns across the eight sites?
Number (%) for whom it was feasible to quantify oral and depots anti-psychotic treatment prescribing in PwID as chlorpromazine equivalent dose values across different healthcare trusts in England and Wales. | Through study completion, an average of 6 months
  Feasibility objective: Is it feasible to quantify anti-psychotic treatment (oral and long-acting IM injectables (depots) prescribing in PwID as chlorpromazine equivalent dose values across different healthcare Trusts in England and Wales?

CONTACTS AND LOCATIONS:
Overall Officials: Professor Shankar, Principal Investigator — University of Plymouth
Locations (8):
- United Kingdom (8):
  - Cheshire and Wirral Partnership NHS Foundation Trust, Chester
  - Coventry and Warwickshire Partnership NHS Trust, Coventry
  - Hertfordshire Partnership University NHS Foundation Trust, Hatfield
  - Leicestershire Partnership NHS Trust, Leicester
  - Central and North West London NHS Foundation Trust, London
  - North East London NHS Foundation Trust, London
  - Cornwall Partnership NHS Foundation Trust, Redruth
  - Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branford D, Shankar R. Antidepressant prescribing for adult people with an intellectual disability living in England. Br J Psychiatry. 2022 Aug;221(2):488-493. doi: 10.1192/bjp.2022.34. PMID 35249557
- [Background] Howkins J, Hassiotis A, Bradley E, Levitas A, Sappok T, Sinai A, Thakur A, Shankar R. International clinician perspectives on pandemic-associated stress in supporting people with intellectual and developmental disabilities. BJPsych Open. 2022 Apr 18;8(3):e84. doi: 10.1192/bjo.2022.49. PMID 35431024
- [Background] Tromans S, Kinney M, Chester V, Alexander R, Roy A, Sander JW, Dudson H, Shankar R. Priority concerns for people with intellectual and developmental disabilities during the COVID-19 pandemic. BJPsych Open. 2020 Oct 29;6(6):e128. doi: 10.1192/bjo.2020.122. PMID 33118913
- [Background] Naqvi D, Perera B, Mitchell S, Sheehan R, Shankar R. COVID-19 pandemic impact on psychotropic prescribing for adults with intellectual disability: an observational study in English specialist community services. BJPsych Open. 2021 Dec 6;8(1):e7. doi: 10.1192/bjo.2021.1064. PMID 34865678
- [Background] Leucht S, Samara M, Heres S, Davis JM. Dose Equivalents for Antipsychotic Drugs: The DDD Method. Schizophr Bull. 2016 Jul;42 Suppl 1(Suppl 1):S90-4. doi: 10.1093/schbul/sbv167. PMID 27460622
- [Background] Patel MX, Arista IA, Taylor M, Barnes TR. How to compare doses of different antipsychotics: a systematic review of methods. Schizophr Res. 2013 Sep;149(1-3):141-8. doi: 10.1016/j.schres.2013.06.030. Epub 2013 Jul 8. PMID 23845387
- [Background] Shankar R, Wilcock M, Deb S, Goodey R, Corson E, Pretorius C, Praed G, Pell A, Vujkovic D, Wilkinson E, Laugharne R, Axby S, Sheehan R, Alexander R. A structured programme to withdraw antipsychotics among adults with intellectual disabilities: The Cornwall experience. J Appl Res Intellect Disabil. 2019 Nov;32(6):1389-1400. doi: 10.1111/jar.12635. Epub 2019 Jun 13. PMID 31192534
- [Background] Mehta H, Glover G. Psychotropic drugs and people with learning disabilities or autism, 2019. Public Health England.
- [Background] National Health Service. Stopping over medication of people with a learning disability, autism or both (STOMP). NHS England " Stopping over medication of people with a learning disability, autism or both (STOMP) [Accessed 15th December 2023).
- [Background] Taylor DM, Barnes TR and Young AH. The Maudsley prescribing guidelines in psychiatry. 13th ed. West Sussex: Wiley-Blackwell; 2018.
- [Background] National Health Service. Statistical process control tool. https://www.england.nhs.uk/statisticalprocess-control-tool/ [Accessed 15th December 2023].
- [Derived] Stanyard E, Neilens H, Allgar V, Bailey M, Musicha C, Purandare K, Perera B, Roy A, Sawhney I, Watkins L, Jaydeokar S, Lennard S, Mitchell S, McGowan P, Laugharne R, Tromans SJ, Shankar R. A novel way to understand and communicate the burden of AntiPsycHotic prescribing for adults across specialist Intellectual Disability services in England and Wales: the APHID feasibility study protocol. Front Health Serv. 2025 May 9;5:1393805. doi: 10.3389/frhs.2025.1393805. eCollection 2025. PMID 40416595